CLINICAL TRIAL: NCT01623492
Title: Eisenmenger Quality Enhancement Research Initiative
Acronym: ES-QuERI
Status: Completed | Type: Observational
Sponsor: Actelion (Industry)
Collaborators: Canadian Heart Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: AC-052-435
Record Dates: First submitted 2012-05-09; First posted 2012-06-20 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Eisenmenger
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Eisenmenger Complex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Blood samples will be collected at Baseline and at each of the annual visits. In addition, urine sampling will be performed at Baseline. An analysis of biomarkers will be performed at a hospital core laboratory.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- diagnosis of Eisenmenger Syndrome: subjects with diagnosis of Eisenmenger Syndrome
  Interventions: Other: Subjects with diagnosis of Eisenmenger Syndrome

INTERVENTIONS:
Other: Subjects with diagnosis of Eisenmenger Syndrome — 1. Antibiotic recommendation for SBE prophylaxis and influenza vaccine
  2. Contraception counseling, and recommendations regarding avoidance of pregnancy
  3. Documentation and prescription of the specific medications:
     1. Oxygen
     2. Diuretic
     3. ASA, Anticoagulant
     4. CCB, BB, ACEI, ARB
     5. Iron Supplementation
     6. Allopurinol
     7. PAH specific therapy
  Other Names: management of Eisenmenger Syndrome

SUMMARY:
Eisenmenger Quality Enhancement Research Initiative (QuERI) is a multi-center, observational, US-based longitudinal program, with enrollment of consecutive Eisenmenger patients who meet enrollment. Patient data will be collected prospectively for three years. Individual physician feedback will be provided on data collected with the purpose of improving the management of patients - quality enhancement research initiative (QuERI) process.

DETAILED DESCRIPTION:
Approximately 200 male and female adult patients with a history of Eisenmenger will be recruited from approximately 50 cardiology practices over a period of 18 months and will be followed up every six months for the period of three years. Consecutive patients in each practice meeting inclusion and exclusion criteria should be considered for the study. Participating sites will be asked to maintain a screening log to identify which inclusion or exclusion criteria was not met thus excluding them from the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Diagnosis of Eisenmenger syndrome based on right heart catheterization data
* Right to Left intra-cardiac shunting
* PAH
* Need for comprehensive management according to guidelines and peer-reviewed evidence
* Ability and desire to execute the consent for follow up

Exclusion Criteria:

* Poor mental function, drug, or substance (e.g.,alcohol) abuse, or unstable psychiatric illness, which, in the opinion of the investigator, may interfere with optimal participation in the study
* Prior inclusion in this program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 adult patients with Eisenmenger Syndrome recruited from approximately 50 US cardiology practices.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Characterization of the clinical course of patients with Eisenmenger Syndrome | up to 3 years
  The management of Eisenmenger Syndrome patients over the three year registry period will be compared with established national guidelines. In addition, The Minnesota Living with Heart Failure questionnaire (MLHFQ) will be collected.

SECONDARY OUTCOMES:
Characterization of the demographics of patients with Eisenmenger Syndrome | baseline (visit 1) thru end of study (3 years)
Identification of clinical predictors of short-term and long-term outcomes of patients with Eisenmenger Syndrome. | baseline (visit 1) thru end of study (3 years)
Characterization of patients treated with PAH-specific medications to patients untreated with PAH-specific medications. | baseline (visit 1) thru end of study (3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Landzberg, MD, Study Chair — Harvard Medical School / Boston Adult Congenital Heart; Gary Palmer, MD, MBA, Study Director — Actelion Pharmaceuticals U.S., Inc.